CLINICAL TRIAL: NCT01886651
Title: The Influence of Thiopurine Methyltransferase Activity on Bone Marrow- and Hepato-toxicity After High-dose Methotrexate in Childhood Acute Lymphoblastic Leukemia
Brief Title: The Influence of Thiopurine Methyltransferase Activity on Toxicity After High-dose Methotrexate in Childhood Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Nordic Society for Pediatric Hematology and Oncology (Other)
Responsible Party: Principal Investigator, Kjeld Schmiegelow, Professor, Rigshospitalet, Denmark
Other Study IDs: NOPHO ALL92 study HDM TPMT
Record Dates: First submitted 2013-06-21; First posted 2013-06-26 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia; child; 6-mercaptopurine; methotrexate
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood stored for a subset of patients
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to explore the impact of thiopurine methyltransferase (TPMT) activity on the risk of HDM-related bone marrow- and hepatotoxicity and treatment interruptions during maintenance therapy for children with ALL.

Hypothesis of the study: Patients with TPMT activity compatible with TPMT low activity polymorphisms have an increased risk of toxicity following high-dose methotrexate (HDM) compared to children with normal TPMT activity.

DETAILED DESCRIPTION:
High-dose methotrexate (HDM) given concurrently with oral 6-mercaptopurine (6MP) may be followed by myelotoxicity, which may necessitate treatment interruption and thus interfere with the efficacy of the treatment of childhood ALL. Several studies have indicated that MTX and 6MP act synergistically. It has previously been reported that the risk of significant bone-marrow suppression is increased if oral 6MP is coadministered with HDM during maintenance therapy and that reductions of the dose of concurrently given oral 6MP can reduce the risk of significant myelotoxicity following HDM. MTX may increase the bioavailability of 6MP through inhibition of xanthine oxidase, which catabolizes 6MP. In addition, MTX may through inhibition of de novo purine synthesis enhance the availability of 6-thioguanine nucleotides (6TGN) that primarily exert the cytotoxic effect of 6MP.

The enzyme TPMT competes with the formation of 6TGN, as it methylates 6MP and thus create relatively non-toxic metabolites. TPMT heterozygous patients with one wild type and one low-activity allele have a higher risk of myelosuppression and treatment interruption compared to patients with TPMT wild type. Furthermore, TPMT heterozygous patients have a reduced risk of relapse and a higher risk of secondary malignancy compared to patients with TPMT wild type.

Little has been published on the influence of both TPMT activity and 6MP dosage on myelo- and hepatotoxicity following HDM.

ELIGIBILITY:
Inclusion Criteria:

* included in the NOPHO ALL92 protocol
* available TPMT phenotype
* treated at least once with HD-MTX 5.0 g/m2 (+- 10%) during maintenance therapy
* at least one available measurement on blood counts or alanine aminotransferase levels 28 days after HD-MTX

Exclusion Criteria:

* HR ALL
* children with Down Syndrome
* Events during maintenance therapy
* TPMT deficiency

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study cohort was based on patients enrolled in the NOPHO ALL92 protocol, where 97% of all eligible patients were included.
  Participation in this study was on the basis of TPMT status that was randomly missing.
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Toxicity of treatment, degree of myelo- and hepatotoxicity | 7-28 days after high-dose methotrexate

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Schmiegelow, M.D., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Kjeld Schmiegelow, Copenhagen, Denmark